CLINICAL TRIAL: NCT06726174
Title: Phase I Clinical Trial of Corneal Endothelial Cell Therapy for Corneal Endothelial Cell Dysfunction
Brief Title: Cell Therapy for Corneal Endothelial Cell Dysfunction
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202304098MINB
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-04

CONDITIONS: Corneal Endothelial Cell Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cell (Experimental)
  Interventions: Drug: ECCEC

INTERVENTIONS:
Drug: ECCEC — 0.5-1x10^6 cells/300 uL, intracameral injection.

SUMMARY:
Culture endothelial cells harvested from donor corneal tissue to treat corneal endothelial cell dysfunction. After ex vivo cultivation, the cells will be injected into anterior chamber and endothelial cells will settle down and adhere to the denuded Descemet's membrane. Eventually, they will reconstitute functional corneal endothelium to subside the corneal edema and improve the visual acuity.

ELIGIBILITY:
Inclusion Criteria:

-

Patient who's one eye or both eyes diagnosed with corneal endothelial cell dysfunction who met the following inclusion criteria were deemed eligible:

1. A BCVA of < 0.5.
2. CECs could not be observed via specular microscopy or CEC density was < 500 cells/mm2.
3. Corneal edema with a corneal thickness > 650 μm.
4. Patient age at the time of obtaining written consent was between 20 and 90 years.
5. Written informed consent could be obtained. If both eyes meet the criteria of a. to c., the treatment eye in this trial will be the one with more sever vision impairment which caused by cornea endothelial cell dysfunction.

Exclusion Criteria:

- Patients who met the following criteria parameters were deemed ineligible and were excluded from the study.

1. Patients with corneal infection (i.e., fungus, bacteria, virus. Etc.).
2. The treatment eye had been cataract surgery, pupilloplasty, or the vision or complication is not stabilized post-operation within one month before transplantation.
3. The treatment eye had received corneal transplantation, other eye surgeries, retinal laser, any kind of invasive eye treatment or drug injection within three months.
4. Pregnant patients (the urine or blood pregnancy test of woman of childbearing potential* is positive) or patients who had recently given birth and were nursing the newborn child.

   *：A woman of childbearing potential (WOCBP) is defined as a premenopausal female capable of becoming pregnant. This includes women on oral, injectable, or mechanical contraception; women who are single; women whose husbands have been vasectomized or whose husbands have received or are utilizing mechanical contraceptive devices.
5. Patients with a hemorrhagic disease (In the patients who is taking Warfarin, the INR is over 3.0.).
6. Patients who were judged by the attending physicians to be incapable of understanding the procedure or of providing sufficient corporation due to mental retardation or mental disorder.
7. Glaucoma patients with poor IOP control (Patients with maximum dosage of glaucoma medicines (Prostaglandin analogue, beta-blocker, alpha2 agonist, and carbonic anhydrase inhibitor) or after surgery, the IOP cannot be controlled under 25 mmHg.).
8. Patients with acute eye infection or inflammation (i.e., bacterial or fungal infection, acute uveitis.)
9. Diabetic patients with a poor blood-sugar control (Patients with HbA1c > 10% within the past three months.).
10. Patients who were hypersensitive to steroids.
11. Patients with systemic autoimmune disease (i.e., systemic lupus erythematosus, Behcet's disease, etc.)
12. Patients strongly suspected to have a severe visual disorder due to concomitant other factors.
13. Patients who had already received this therapy.
14. Patients who had used or were planning to use an anti-cancer drug.
15. Patients with a past history of heart disease (i.e., myocardial infarction, heart failure, severe arrhythmia, etc.) or a cerebral vascular disorder.
16. Patients for whom it has been determined by the principal investigator or other co-investigators that there will be complications with the patient participating in the study for other reasons.
17. Patients who are allergic to the drug or ingredients used in this trial.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
CEC density | 24-weeks
  > 500 cells/mm2

SECONDARY OUTCOMES:
Corneal thickness | 24-weeks
  < 650 μm

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan